CLINICAL TRIAL: NCT02582229
Title: A Prospective Study to Evaluate the Efficacy of an Endoluminal-suturing Device (Endomina TM) as an Aid for Endoscopic Gastric Reduction.
Acronym: Endomina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2015/432
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventionnal (Experimental): The intervention will be performed under general anesthesia with tracheal intubation. Endomina will be introduced into the stomach over guide wires and then fixed to the endoscope. The procedure will include the placement of 4-6 transmural anterior-posterior sutures after argon plasma coagulation of the tissue opposition areas in order to ensure persistence of the pouch reduction. Patient will be kept overnight after the procedure.
  Interventions: Device: Endomina

INTERVENTIONS:
Device: Endomina — The intervention will be performed under general anesthesia with tracheal intubation. Endomina will be introduced into the stomach over guide wires and then fixed to the endoscope. The procedure will include the placement of 4-6 transmural anterior-posterior sutures after argon plasma coagulation of the tissue opposition areas in order to ensure persistence of the pouch reduction. Patient will be kept overnight after the procedure.

SUMMARY:
Surgery is the only effective treatment for morbid obesity and can be divided into restrictive surgeries (Lap Band and Sleeve gastrectomy), malabsorptive surgeries (Biliary pancreatic deviation and duodenal switch) or a combination of both (RYGBP).

This later technique is the most common and most effective surgical procedure performed worldwide and has been processed to be an effective treatment of morbid obesity and its complications, achieving excess weight loss of 65 to 80 % ; 1-2 years after surgery (1,2).

Vertical gastric plication is a novel surgical approach for reducing the stomach capacity. Anterior surface plication and greater curvature plication are variations of vertical gastric plication that reduce the gastric capacity through infolding of the anterior surface or greater curvature of the stomach, respectively. These approaches have been tested, with positive results (3,4).

A transoral or endoluminal approach (ie, a procedure that requires no incision, because access is granted through the mouth) offers the potential for additional benefit to the patient, because the procedures continue to become more and more minimally invasive.

Advances in endoluminal devices are now allowing clinicians the ability to begin exploring bariatric procedures performed via flexible endoscopy. Although these procedures may not be as effective as their surgical counterparts, these less-invasive options may relieve patients of the significant risks associated with surgery (5).

DETAILED DESCRIPTION:
Endomina (Endo Tools Therapeutics, Nivelles, Belgium) is CE mark robot driven device that may be attached to an endoscope inside the body and allows remote manipulation of the arms of devices during a peroral intervention. It offers the possibilities of making transoral surgical full thickness sutures and may allow performing, via a transoral route.

After a first trial on pigs (safety) we did a second trial on human. This trial included 11 patients treated with the same technique. There were no complications and the short term results were encouraging.

Study design:

Prospective, non-randomized, interventional, open-label, multi-center efficacy study.

Objectives:

Study to evaluate the efficacy of an endoluminal vertical gastroplasty (EVG) using an endoluminal-suturing device. In the literature the efficacy of an endoluminal technique is defined as a loss of weight of 25% excess weight loss (EWL) sustained at 1 year (6).

Endpoints Secondary endpoint: Efficacy Information on efficacy will be obtained by measurements of total weight loss and excess weight loss during 12 months Secondary endpoint: Safety Safety will be characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants.

In addition, safety assessments will be determined based on physical examination (vital signs) and laboratory tests during scheduled visits. Safety evaluations will also be performed to ensure no subsequent adverse events have occurred and to ensure any adverse events during the trial that are considered on-going are stable or have resolved. Safety will be assessed at 1, 3, 6 and 12 months following the intervention.

Sample size •40 patients will be enrolled Based on the result of our previous study, with a beta power of 80% and an alpha error of 5%, the number of patient needed to detect a 25% EWL reduction at one year is 34. Considering a lost to follow-up of 10%, 40 patients is required.

Study duration:

•6 months of enrolment and 12 months of follow up Overall design This will be a prospective, non-randomized, open-label, multi-center, interventional, efficacy study.

A period of approximately 6 months is anticipated form the time the first patient is enrolled to the completion of the last patient. There will be no randomization in this study.

Once baseline eligibility criteria have been met all patients will undergo the same treatment protocol. A subject will be considered "enrolled" if he/she has signed the informed consent, passed all screening criteria and has undergone a procedure.

Criteria for discontinuation If a subject discontinues participation in the study, he or she will be contacted in order to obtain information about the reason(s) for discontinuation and collection of any potential AEs. The Investigator will document the reason for Subject Withdrawal on the Patient Case Report Form (CRF). Discontinued patients will be followed until all AEs resolve or until the Investigator decides that follow-up are no longer necessary.

Study Design:

Devices used during the protocol In addition to Endomina device (provided as companionate by Endotools Options) any other required endoscopic accessories can be used during the procedure.

Point of enrollment A subject will be considered "enrolled" if he/she has signed the informed consent, passed all screening criteria and has agreed to the procedure.

Study duration and number of subjects A period of approximately 6 months is anticipated form the time the time the first patient is enrolled to the completion of the last patient.

Lab tests and other screening procedures can occur as early as 30 days prior to scheduled procedure.

The participants will be followed as follow:

* Day (-1): Admission
* Day (0): Procedure
* Day (+1): Clinical Follow up and discharge (i.e. if no adverse effects observed)
* 1 month: Clinical assessment
* 3 month: Follow up endoscopy, Clinical assessment
* 6 month: Clinical assessment
* 12 month: Clinical and endoscopic assessment On Parallel a nutritional specialist will monitor the patient on quarterly basis (1,3,6,12).

Study procedures The intervention will be performed under general anesthesia with tracheal intubation. Endomina will be introduced into the stomach over guide wires and then fixed to the endoscope. The procedure will include the placement of 4-6 transmural anterior-posterior sutures after argon plasma coagulation of the tissue opposition areas in order to ensure persistence of the pouch reduction. Patient will be kept overnight after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21-64 years;
2. BMI between 30 to 40 kg/m²
3. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment, endoscopy, radiography, as well as laboratory investigations.
4. Must be able to understand and be willing to provide written informed consent.

Exclusion Criteria:

1. Achalasia and any other esophageal motility disorders
2. Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity.
3. Hypertension: uncontrolled hypertension during last 3 month
4. Severe renal, hepatic, pulmonary disease or cancer;
5. GI stenosis or obstruction
6. Pregnancy or breastfeeding
7. Impending gastric surgery 60 days post intervention;
8. Currently participating in other study

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Weight Loss | one year
  Weight loss - Excess Weight Loss - BMI

SECONDARY OUTCOMES:
Complications | one year
  Vital signs - Pain - Bleeding - Perforation - other

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Deviere, MD,PhD, Study Director — Hopital Erasme, Gastroenterology Department
Locations (3):
- Gastroenterology Department Erasme Hospital, Brussels, Belgium
- Internal cilic - department of Gastroenterology - University Hospital, Ostrava, Czechia
- U.O. Endoscopia Digestiva Chirurgica, Roma, Italy

REFERENCES:
- [Result] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Result] Magro DO, Geloneze B, Delfini R, Pareja BC, Callejas F, Pareja JC. Long-term weight regain after gastric bypass: a 5-year prospective study. Obes Surg. 2008 Jun;18(6):648-51. doi: 10.1007/s11695-007-9265-1. Epub 2008 Apr 8. PMID 18392907
- [Result] Fogel R, De Fogel J, Bonilla Y, De La Fuente R. Clinical experience of transoral suturing for an endoluminal vertical gastroplasty: 1-year follow-up in 64 patients. Gastrointest Endosc. 2008 Jul;68(1):51-8. doi: 10.1016/j.gie.2007.10.061. Epub 2008 Mar 19. PMID 18355825
- [Result] Paxton JH, Matthews JB. The cost effectiveness of laparoscopic versus open gastric bypass surgery. Obes Surg. 2005 Jan;15(1):24-34. doi: 10.1381/0960892052993477. PMID 15760496
- [Derived] Huberty V, Machytka E, Boskoski I, Barea M, Costamagna G, Deviere J. Endoscopic gastric reduction with an endoluminal suturing device: a multicenter prospective trial with 1-year follow-up. Endoscopy. 2018 Dec;50(12):1156-1162. doi: 10.1055/a-0630-1224. Epub 2018 Jun 15. PMID 29906810